CLINICAL TRIAL: NCT00395031
Title: The Effects of Ziprasidone 320 mg on Glucose and Plasma Lipids in Patients With Diabetes Type II and Schizophrenia or Schizoaffective Disorder
Brief Title: Effect of Ziprasidone on Glucose & Plasma Lipids in Diabetes (II) and Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Manhattan Psychiatric Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Jean-Pierre Lindenmayer, Director of Psychopharmacology Research, Manhattan Psychiatric Center, NY, RFMH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03I/C24; Pfizer Reference # 2001-0448 (Other Grant/Funding Number: Pfizer Inc)
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; Schizoaffective Disorder; metabolic markers; ziprasidone; diabetes
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Diabetes Mellitus | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ziprasidone (Other): Open label
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — Ziprasidone dose of between 40 mg po bid to 160 mg po bid for 8 weeks
  Other Names: Geodon

SUMMARY:
The aim of the protocol is to study the effects of 320 mg/day of ziprasidone (Geodon) on glucose and lipid metabolism of patients with both Diabetes Type II (DM) and schizophrenia or schizoaffective disorder, after switching their antipsychotic medication/s from typical and/or atypical to ziprasidone monotherapy.

DETAILED DESCRIPTION:
Inpatients with DSM IV diagnosis of schizophrenia or schizoaffective disorder and DM II will be enrolled after giving informed consent. Participants may stay on their original ward at MPC, if their clinical care would be better served on their home ward because of patient programs and/or continuity of care reasons. Patients recruited from other participating sites will be transferred to MPC research ward.

There will be a screening phase (two weeks) on the prior antipsychotic regimen, a cross-titration phase (three week) and a ziprasidone phase (eight weeks; four time points).

All medications, except for the antipsychotic agents, will be kept stable throughout the protocol. These medications may include anticholinergics, mood stabilizers and antidepressants. After the screening phase lasting two weeks, patients will enter the cross-titration phase lasting three week. The cross titration schedule will be changed in accordance with Deutschman & Deutschman's 2005 recommendations. The current antipsychotic will be gradually decreased to zero and ziprasidone will be started at 40 mg bid po and raised up to 160 mg po bid during the cross-titration phase, according to clinical response and tolerance. After the cross-titration phase has concluded, the ziprasidone dose will range from 80 mg bid p.o. to 160 mg bid p.o. daily according to clinical response during the eight week treatment phase.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years
2. DSM IV diagnosis of schizophrenia (all subtypes) or schizoaffective disorder
3. Diabetes Mellitus type II treated with oral antidiabetic drugs or insulin
4. Stable dose of antipsychotic regimen for previous one month.
5. Stable dose of antidepressant regimen for previous one month.
6. Stable dose of adjunctive mood stabilizer and/or anticholinergic regimen for previous 1 month
7. Signed informed consent
8. Absence of significant cardiovascular pathology as demonstrated by EKG (QTc < 450 millisec)
9. Absence of severe medical conditions (except for DM) requiring frequent changes in medication.

Exclusion Criteria:

1. DSM IV diagnosis other than Schizophrenia or Schizoaffective disorder
2. Unstable epilepsy
3. Acute, unstable or significant medical condition
4. Suicidal or physically violent behavioral episodes in the previous month
5. Current DSM IV diagnosis of substance or alcohol abuse with positive urine toxicology in the past two weeks.
6. Liver enzyme test values ≥ three times upper normal limit for AST, ALT, GGT, and Alkaline Phosphatase; ≥ two times upper limit for LDH.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2003-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Reduced Glucose, Cholesterol and Lipid Levels | 11 weeks

SECONDARY OUTCOMES:
Reduction in dose requirement for antiglycemic agents | 11 week
Improvement in quality of life & Positive and Negative Symptoms | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Kaushik, M.D., Study Chair — Manhattan Psychiatric Center, New York University, Nathan Kline Institute; Jean-Pierre Lindenmayer, M.D., Principal Investigator — Manhattan Psychiatric Center, New York University, Nathan Kline Institute
Locations (1):
- Manhattan Psychiatric Center, New York, New York, United States

REFERENCES:
- [Background] Levy WO, Robichaux-Keene NR, Nunez C. No significant QTc interval changes with high-dose ziprasidone: a case series. J Psychiatr Pract. 2004 Jul;10(4):227-32. doi: 10.1097/00131746-200407000-00003. PMID 15552544
- [Background] Deutschman DA, Deutschman DH. High-dose ziprasidone in treatment-resistant schizophrenia and affective spectrum disorders: a case series. J Clin Psychopharmacol. 2007 Oct;27(5):513-4. doi: 10.1097/JCP.0b013e31814cface. No abstract available. PMID 17873687
- [Derived] Kaushik S, Maccabee N, Kaushik S, Lindenmayer JP. Activation induced by high-dose ziprasidone: a case report. J Clin Psychiatry. 2009 Sep;70(9):1326-7. doi: 10.4088/JCP.08l04400. No abstract available. PMID 19818257
- See also: Site dedicated exclusively to ziprasidone sponsored by PharmaPromo a division of Anakena Internet Services. — http://www.ziprasidone.com/
- See also: Ziprasidone information on medlineplus, a service of NIH — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a699062.html